CLINICAL TRIAL: NCT05868200
Title: Anti-Inflammatory Efficacy of Ginger Containing Dentifrice in the Control of Biofilm Induced Gingivitis: a 3 Months Randomized Parallel Clinical Trial
Brief Title: Anti-Inflammatory Efficacy of Ginger Containing Dentifrice in the Control of Biofilm Induced Gingivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Zainab Zuhair Alalawi, Principal Investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 523622
Record Dates: First submitted 2023-04-16; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — hydrated silica gel-based toothpaste

STUDY DESIGN:
Intervention Model Description: 80 subjects with plaque induced gingivitis, caused by accumulation of plaque, will be selected and enrolled in this study. Subsequently, subjects will be equally divided and randomly allocated for two groups, each group received a similar number of subjects (n=40) with a 1:1 allocation.
Who Masked: Participant, Investigator
Masking Description: The products will be packaged in such a way that they are not recognizable neither by the operator, nor by the patient. Each package will be assigned a number that in turn will refer to the type of the product. The association between the number and type of the product will be collected by another operator according to the association carried out by a dedicated software. The operator who will deliver the product will be informed about the type only at the end of the treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capitano zenzero toothpaste (Experimental): Participants will be given the test interventions, Capitano zenzero toothpaste, and will be asked to brushing teeth with this product for two minutes twice per day and will be instructed to refrain from eating and drinking for 30 min after rinsing.
  Interventions: Drug: Capitano zenzero toothpaste
- Colgate total toothpaste (Active Comparator): Participants will be given the test interventions, Colgate total toothpaste, and will be asked to brushing teeth with this product for two minutes twice per day and will be instructed to refrain from eating and drinking for 30 min after rinsing.
  Interventions: Drug: Colgate total toothpaste

INTERVENTIONS:
Drug: Capitano zenzero toothpaste — Filming toothpate formulation, enriched with 3%ginger as active ingredient and Zinc coco sulfate as surfactant, cleansing and emulsifying agent.
  Subjectswill then be given the test intervention, Capitano zenzero toothpaste, and will be asked to brush with it for two minute twice per day and will be instructed torefrain from eating and drinking for 30 min after brushing. participants will be received a toothbrush with medium-hardness bristles .the bass technique method of brushing by was comprehensively explained to all participants.. Next, the participants will be re-evaluated after 3 months .
  Other Names: Ginger toothpaste
  Arms: Capitano zenzero toothpaste
Drug: Colgate total toothpaste — Subjects will then be given Colgate total toothpaste, as an active comparator, and will be asked to brush with it for two minutes twice per day and will be instructed to refrain from eating and drinking for 30 min after rinsing. participants will be received a toothbrush with medium-hardness bristles . participants will be received a toothbrush with medium-hardness bristles .the bass technique method of brushing by was comprehensively explained to all participants.. Next, the participants will be re-evaluated after 3 months .
  Arms: Colgate total toothpaste

SUMMARY:
The goal of this clinical trial is to test efficiency of using toothpaste containing (Ginger) over a period of three month to control on gingival inflammation and plaque accumulation through measuring the clinical periodontal parameters (Gingival Index (GI), Bleeding on probing (BOP) and modified Quigley-Hein Plaque Index (mQHPI ) in comparison with Colgate total toothpastes in patients with biofilm induced gingivitis.

DETAILED DESCRIPTION:
Objectives:

1. Measuring the clinical periodontal parameter (gingival index) and salivary cytokine IL-1β and superoxide dismutase SOD over a period 3 months before and after using Capitano (ginger containing) and Colgate total toothpastes for patients with gingivitis.
2. Measuring the clinical periodontal parameter ((Gingival Index (GI), Bleeding on probing (BOP) and modified Quigley-HeinPlaque Index (mQHPI )) over a period 3 months before and after using Capitano (ginger containing) and Colgate total toothpastes for patients with gingivitis by ELISA.
3. correlation between ( Interleukin 1 beta and SOD) and clinical periodontal parameters

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 20-35 who will volunteer to participate.
2. Apparently good general health.
3. Patients with gingivitis (having ≥30% bleeding sites with no PPD >3 mm, intact periodontium and no loss of periodontal attachment).
4. Those with a minimum of 20 natural teeth.

Exclusion Criteria:

* 1. Those with chronic disease, immunocompromised patients, pregnant, on contraceptive and lactating women.

  2. Those currently using any mouthwash. 3. Those on antibiotic therapy and anti-inflammatory medications during the study and at the last 2 months before the study.

  4. Those having a history of hypersensitivity to any product used in the present study.

  5. Those with a recent tooth extraction. 6. Those having periodontitis. 7. Those who smoker or alcoholism. 8. Those with extensive untreated dental caries, diseases of hard and soft palate and subjects wearing orthodontic appliances, removable dentures, implant, crown and bridge or presenting with abnormal salivary flow.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-02-12 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Change in Gingival index | 0 ,3 months
  Subjects will undergo the measurement of gingival index according to Loe & Silness, designed to assess the severity and quality of gingival inflammation in an individual or population. The gingival inflammation is assessed on the basis of color, consistency and bleeding on probing. The gingiva surrounding the tooth is assessed at four sites: mesio-facial papilla, facial marginal gingiva, disto-facial papilla and lingual marginal gingiva. Data will be collected based on four possible clinical conditions:
  0=Normal gingiva1=Mild Inflammation-Slight change in color, Slight odema. No bleeding on probing2=Moderate inflammation-redness,odema and glazing. Bleeding on probing 3=Sever inflammation-marked redness and edema.Ulceration.Tendency to spontaneous bleeding.
Mean relative changes in Interleukin 1 beta level in salivary Fluid. | 0 ,3 months
  Mean relative changes in Interleukin 1 beta level in salivary fluid after brushing with different comparators from baseline at 3 months.
Mean relative changes in superoxide dismutase SOD level in salivary Fluid. | 0 ,3 months
  Mean relative changes in superoxide dismutase SOD level in salivary fluid after brushing with different comparators from baseline at 3 months.

SECONDARY OUTCOMES:
Changes in BOP score | 0 ,3 months
  For recording BOP score, the periodontal probe was inserted with gentle force into the sulcus/pocket until minimal resistance was felt. The probing force presumably was ranging between 20 to 25g. The examination started from the distal surface of the right upper 7 moving mesially to measure all the existing teeth. For each tooth, 6 surfaces were examined; the surface that displayed bleeding on probing was scored 1 and the surface with no bleeding was scored 0
Mean amount plaque between different comparators. | 0 ,3 months
  Mean amount plaque between different comparators as anti-plaque agent after brushing with different comparators using means of modified quigely hein plaque index[ Turesky ,1970]

CONTACTS AND LOCATIONS:
Overall Officials: zainab Al ALawi, H. diploma, Principal Investigator — University of Baghdad
Locations (1):
- Zainab, Baghdad, Iraq